CLINICAL TRIAL: NCT04772326
Title: Impact of Containment and the Current Epidemic on the Sexual Risk-taking of People Using PrEP to Prevent HIV Infection.
Acronym: CoroPrEP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH_2020_10
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: PREP
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PrEP patients undergoing follow-up at Tourcoing hospital
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
People using PrEP to prevent HIV infection have sexual risk-taking behaviors that motivated the prescription of PrEP. Both containment and the current epidemic may affect the sexual behavior of people using PrEP and the risk of acquiring STIs.

Hypotheses regarding the impact of the current epidemic-motivated confinement and its gradual lifting are as follows:

* A decrease in sexual risk-taking during the confinement period, followed by an increase when the confinement is lifted.
* An increase in sexual violence and the use of psychoactive substances.
* An impact on PrEP monitoring and compliance.
* An increase in the incidence of STIs when the confinement is lifted.

ELIGIBILITY:
Inclusion Criteria:

* People using PrEP for HIV prevention being followed up at Tourcoing hospital
* Having given their consent to participate in this study
* Beneficiary of a social insurance plan or entitled person

Exclusion Criteria:

* Minor patient
* Refusal to participate
* Trusteeship
* Curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in all persons using PrEP as prevention against HIV infection undergoing follow-up at Tourcoing Hospital and receiving counseling during months of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Impact of the current epidemic on sexual risk taking of Prep users in the number of partners per month | At day 1
Impact of the current epidemic on sexual risk taking of Prep users in the number of sexual encounters per month | At day 1
Impact of the current epidemic on sexual risk taking of Prep users in the frequency of condom use during anal intercourse | At day 1

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Meybeck, MD, Principal Investigator — CH TOURCOING
Locations (1):
- CH Tourcoing, Tourcoing, France